CLINICAL TRIAL: NCT04751461
Title: CSD210202: An Unblinded, Randomized, Crossover, Confinement Study to Assess Nicotine Uptake From Electronic Nicotine Delivery Systems
Brief Title: CSD210202: A Study to Assess Nicotine Uptake From Electronic Nicotine Delivery Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSD210202
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Smoking; Smoking Behaviors; Tobacco Use; Tobacco Smoking
MeSH Terms: conditions — Smoking; Tobacco Use; Tobacco Smoking | interventions — HTR3D protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Product usage order ABECD (Experimental): Subjects will use each of the 5 products (ABECD) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order BCADE (Experimental): Subjects will use each of the 5 products (BCADE) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order CDBEA (Experimental): Subjects will use each of the 5 products (CDBEA) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order DECAB (Experimental): Subjects will use each of the 5 products (DECAB) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order EADBC (Experimental): Subjects will use each of the 5 products (EADBC) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order DCEBA (Experimental): Subjects will use each of the 5 products (DCEBA) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order EDACB (Experimental): Subjects will use each of the 5 products (EDACB) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order AEBDC (Experimental): Subjects will use each of the 5 products (AEBDC) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order BACED (Experimental): Subjects will use each of the 5 products (BACED) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order CBDAE (Experimental): Subjects will use each of the 5 products (CBDAE) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E

INTERVENTIONS:
Other: Product A — P0213420, a 1.8% nicotine ENDS product
Other: Product B — P0213520, a 1.8% nicotine ENDS product
Other: Product C — P0211220, a 1.8% nicotine ENDS product
Other: Product D — P0211820, a 1.8% nicotine ENDS product
Other: Product E — P0213417, a 2.4% nicotine ENDS product

SUMMARY:
This is an open-label, randomized, 5-way crossover study designed to evaluate plasma nicotine pharmacokinetic (PK) parameters following an ad libitum use of Electronic Nicotine Delivery System (ENDS) investigational products (IPs) in a confinement setting by generally healthy combustible cigarette (CC) smokers.

DETAILED DESCRIPTION:
Potential subjects will complete a pre-screening interview and a Screening Visit to assess their eligibility within 45 days prior to enrollment, randomization and confinement.

Following the Screening Visit, eligible subjects will be scheduled for a check-in and randomization visit. At the check-in and randomization visit, subjects' continued eligibility will be confirmed prior to being randomized to a product use sequence and beginning their 6 nights and 7 days of confinement.

Starting on study Day 1, subject will start a Pre-study ENDS IP Acclimation Period through Day 2. Subjects will be asked to acclimate to each of the ENDS IP at least once, while having access to their usual brand (UB) cigarettes for ad libitum use. Starting on Day 3, subjects will participate in five separate Test Sessions for nicotine PK assessment, one for each ENDS IP. For approximately a half day prior to each respective Test Session (starting on Day 2), subjects will use their assigned ENDS IP for the following day's Test Session at least twice.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
2. Generally healthy male or female, 21 to 60 years of age, inclusive, at the time of consent.
3. Expired breath carbon monoxide level is ≥ 10 ppm and ≤ 100 ppm at Screening.
4. Positive urine cotinine test at Screening.
5. Smokes only filtered, menthol or non-menthol combustible cigarettes, 83 mm to 100 mm in length.
6. Agrees to smoke same UB combustible cigarette throughout the study period. UB combustible cigarette is defined as the cigarette brand style currently smoked most frequently by the subject.
7. Smokes at least 10 cigarettes per day (on average) and inhales the smoke, for at least 6 months prior to Screening. Brief periods of abstinence due to illness, quit attempt (prior to 30 days of Screening), or clinical study participation (prior to 30 days of Screening) will be allowed at the discretion of the Principal Investigator (PI).
8. Willing to use only UB combustible cigarette and ENDS during the study period.
9. Willing to abstain from tobacco and nicotine use for at least 12 hours prior to each Test Session.
10. Females must be willing to use a form of contraception acceptable to the PI from the time of signing informed consent until End-of-Study.
11. Agrees to in-clinic confinement of 7 days and 6 nights.

Exclusion Criteria:

1. Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI, makes the study subject unsuitable to participate in this clinical study.
2. History, presence of, or clinical laboratory test results indicating diabetes.
3. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95mmHg, measured after being seated for five minutes.
4. Weight of ≤ 110 pounds.
5. Hemoglobin level is < 12.5 for females or <13.0 for males g/dL at Screening.
6. Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening Visit. As-needed treatment, such as inhalers, may be included at the PI's discretion pending approval from the Medical Monitor.
7. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
8. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
9. Use of an ENDS or tobacco or nicotine-containing products other than cigarettes (e.g., lozenges, moist snuff) within (≤) 30 days prior to Screening.
10. Use of any medication or substance that aids in smoking cessation, including but not limited to any NRT (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to the signing of informed consent.
11. History or presence of bleeding or clotting disorders.
12. Any use of anticoagulants or aspirin (≥ 325 mg/day).
13. Whole blood donation within 8 weeks (≤ 56 days) prior to the signing of informed consent.
14. Plasma donation within (≤) 7 days prior to the signing of informed consent.
15. Plans to donate whole blood or plasma prior to Enrollment and Study Day 1.
16. Participation in another clinical trial within (≤) 30 days prior to the signing of informed consent. The 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing the ICF in the current study.
17. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
18. Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
19. A positive urine drug screen without evidence of prescribed corresponding concomitant medication(s) at Screening or Day 1.
20. Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or a previous attempt within (≤) 30 days prior to the signing of the ICF.
21. Drinks more than 21 servings of alcoholic beverages per week or has a positive alcohol breathalyzer result at Screening or Day 1.
22. Employed by a tobacco or nicotine company, the study site, or handles tobacco- or nicotine-containing products as part of their job.
23. Determined by the PI to be inappropriate for this study. *Subjects will be advised against scheduling of whole blood or plasma donation following study completion for at least 7 days.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
AUCnic0-240 | 0 to 240 minutes
  Baseline-adjusted area under the plasma nicotine concentration-versus-time curve from time zero to 240 minutes after the start of IP use
Cmax | 240 minutes
  Maximum baseline-adjusted plasma concentration of nicotine

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hong, MD, Study Director — RAIS
Locations (1):
- AMR Knoxville, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No